CLINICAL TRIAL: NCT02643264
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) of the Insula for Treatment of Alcohol Addiction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Markus Heilig, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIU2015/130-31
Record Dates: First submitted 2015-12-21; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Alcohol Addiction
Keywords: insula; alcohol addiction; transcranial magnetic stimulation
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rTMS 10 Hz (Experimental): Deep Repetitive Transcranial Magnetic Stimulation (rTMS, 10 Hz) of the insula ,15 stimulation sessions (1 daily, 5 days / week).
  Interventions: Other: rTMS 10 Hz targeting the insula
- rTMS Sham (Sham Comparator): Sham Repetitive Transcranial Magnetic Stimulation (rTMS, Sham),15 stimulation sessions (1 daily, 5 days / week).
  Interventions: Other: Sham rTMS

INTERVENTIONS:
Other: rTMS 10 Hz targeting the insula — Participants will receive a total of 15 sessions of rTMS targeting the insula bilaterally, Stimulation will be delivered at an intensity of 120% of the motor threshold (MT), with a frequency of 10 Hz, delivered as 50 trains of 30 pulses delivered in each train of 3 seconds duration, with a 20 seconds inter-train interval, for a total of 1500 pulses delivered over app. 20 min. On the very first two sessions stimulations will be given at lower strength for adaptation, starting at 100% for the first and 110% for the second session
  Arms: rTMS 10 Hz
Other: Sham rTMS — Sham stimulation with the same regimen as active treatment
  Arms: rTMS Sham

SUMMARY:
The purpose of this study is to investigate the effects of repetitive transcranial magnetic stimulation (rTMS) targeting the insula on alcohol use and neural responses in alcohol-dependent patients.

DETAILED DESCRIPTION:
Objectives: To investigate the effects of repetitive transcranial magnetic stimulation (rTMS) targeting the insula on alcohol use and neural responses in alcohol-dependent patients.

Study population: Treatment seeking alcohol dependent subjects (N=82), aged 18-65 years, who have first completed standard alcohol withdrawal treatment if needed.

Design: This is a double-blind, sham-controlled randomized study, comprising three phases. Participants will be hospitalized during the first two of these, and will be outpatients during the third. During Phase 1 the study (screening; up to 14 days), participants will undergo a set of baseline assessments; this phase will conclude with consent, inclusion and randomization. During Phase 2 (treatment; appr. 3 weeks, with at least the first week being hospitalized), participants will first undergo an MRI scan to collect resting state and structural data, and will then receive one of two treatments: Active (10Hz) rTMS; or sham stimulation, both targeting the insula bilaterally. rTMS sessions will be conducted five times per week, for 3 weeks, for a total of 15 sessions. Stimulation will be with an H-coil designed to reach deeper structures such as the insula. A second MRI scan will be obtained at the end of this phase to assess changes in resting state connectivity, and to evaluate insula activity in tasks known to activate this structure. In addition, a lumbar puncture will be carried out at the end of this phase to assess possible effects on central neurotransmitter and growth factor levels, as indexed in the cerebrospinal fluid. For Phase 3 (follow-up, lasting 12 weeks), patients will be followed as outpatients for 12 weeks, with clinic visits at weeks 1, 2, 4, 8 and 12 post discharge; measures of alcohol use will be collected during this phase.

Outcome measures: The co-primary outcome measures will be heavy alcohol consumption during the follow-up phase, assessed using time-line follow-back methodology; and insula BOLD functional magnetic resonance imaging (fMRI) responses during tasks known to induce insula activation. A number of secondary and exploratory measures will also be assessed, including objective biomarkers of alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 65
2. Current Diagnostic and Statistical Manual (DSM-IV-TR) diagnosis of alcohol dependence
3. Alcohol use in the past month
4. Right handed (self-report)
5. If female, negative urine pregnancy test
6. If female, must either agree to practice an effective birth control method; have a partner with a vasectomy; agree to abstinence from intercourse; be surgically sterile or postmenopausal for at least one year

Exclusion Criteria:

1. Currently pregnant or breastfeeding
2. More than mild cognitive impairment, as determined by a score on the Mini Mental State Examination (MMSE) <24.
3. Current DSM-IV diagnosis of schizophrenia, bipolar disorder, or other psychotic disorder
4. Use in the past 4 weeks of any medication or illicit drug listed as being associated with "a strong potential hazard for application of rTMS due to their significant seizure threshold lowering potential" by the international consensus guidelines for delivery of TMS [104], as self-reported, or detected using urine toxicology screening
5. Any history of clinically significant neurological disorders, including organic brain disease, epilepsy, stroke, brain lesions, multiple sclerosis, previous neurosurgery or personal history of head trauma that resulted in loss of consciousness for > 5 minutes and retrograde amnesia for > 30 minutes (self-reported history).
6. Any history of seizures other than febrile childhood seizures (self-reported history)
7. Signs of increased intracranial pressure as determined by the structural MRI-scan
8. Clinically significant hearing impairment or tinnitus
9. Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head (pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments) or fear of enclosed spaces. Eligibility will be determined by the "MRI Safety Screening Questionnaire" (see Appendix 1) and verified, if necessary, by a radiology consultant.
10. Cannot recline comfortably flat on his/her back for up to 2 hours in the MRI scanner.
11. Any psychiatric, medical or social condition whether or not listed above, due to which, in the judgment of the investigators and after any consults if indicated, participation in the study is not in the best interest of the patient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Heavy Drinking | 12 weeks follow-up from treatment completion
  Reduction in heavy alcohol use during the outpatient follow-up phase (%heavy drinking days) measured by standard Time-Line Follow-Back methodology
Insula activity | Within 5 days of treatment completion
  Insula activity (%signal change, as measured by fMRI BOLD), during a task known to be associated with insula responses, risky decision making

SECONDARY OUTCOMES:
BOLD responses in a battery of standard fMRI tasks that probe processing of alcohol-associated cues, reward function, and emotional responses. | Within 5 days after the last TMS session
Alterations in resting-state connectivity of the insula with other nodes in the putative Salience Network (SN), executive control network (ECN) and the default-mode network (DMN) by rTMS. | Within 5 days after the last TMS session
Objective biomarkers of alcohol use | 12 weeks follow-up from treatment completion
  Gamma-glutamyl transferase (GGT); carbohydrate deficient transferrin (CDT); ethyl glucuronide (EtG) in urine and hair.
Alcohol craving and psychiatric symptoms | 12 weeks follow-up from treatment completion
  Measured by the Penn Alcohol Craving Scale (PACS), mood and anxiety symptoms, as measured using the respective subscales of the Comprehensive Psychiatric Rating Scale (CPRS) and Clinical Global Impression (CGI).
Smoking | 12 weeks follow-up from treatment completion
  Measured by urine cotinine / creatinine ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Markus A Heilig, MD PhD, Principal Investigator — Linkoeping University
Locations (1):
- Linkoping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Yes